CLINICAL TRIAL: NCT01610102
Title: Clinical Performance and Angiographic Results of Coronary Stenting With Absorbable Metal Stents, Clinical Long Term Follow-Up
Brief Title: PROGRESS-AMS 1.0 Clinical Long Term Follow-Up
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1104
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Long Term Safety of the AMS 1.0
Keywords: clinical follow-up; up to 7 years; all patients enrolled in the main study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to collect long term clinical follow-up data on all patients enrolled in the PROGRESS AMS-1.0 study to assess long term safety of the AMS-1.0

DETAILED DESCRIPTION:
The first clinical experience with AMS was in infrapopliteal arteries and demonstrated safety and acceptable patency rates up to 12 months post implantation. These encouraging results led to the initiation of the first trial to treat human coronary lesions with AMS named Clinical Performance and angiographic Results of Coronary Stenting with Absorbable Metal Stents (PROGRESS AMS-1). Although an ischemic driven target lesion revascularization rate of 26.7% (16/60) was observed during the PROGRESS AMS-1 study, it demonstrated that biodegradable magnesium stents can be implanted safely in coronary arteries, and the stents degraded as intended without causing stent thrombosis, myocardial infarction or death at one year. No adverse device effects from the absorbable nature of the stents or its constituents were detected. The continued clinical follow-up and retrospective evaluation of all angiographies and IVUS films on all eligible patients enrolled in the PROGRESS-AMS 1.0 will give important information on the long term safety of absorbable metal scaffolds and thus can support improvement of the device.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form available prior to clinical long term follow-up

Exclusion Criteria:

* Patent did not sign the informed consent form prior to clinical long term follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 63 eligible patints previously enrolled in the PROGRESS AMS-1 study
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | up to 7 years follow-up
  Composite of cardiac death, target vessel myocardial infarction, clinically driven target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Erbel, Prof., Principal Investigator — Westdeutsches Herzzentrum Essen; Esther Gerteis, Study Director — Biotronik AG
Locations (6):
- Austin & Repatriation Medical Centre, Heidelberg, Victoria, Australia
- O.L.V. Ziekenhuis Aalst, Aalst, Belgium
- Westdeutsches Herzzentrum Essen, Essen, North Rhine-Westphalia, Germany
- Catharina Zieckenhuis, Eindhoven, Netherlands
- Switzerland (2):
  - Luzerner Kantonsspital, Lucerne
  - University Hospital Zürich, Zurich